CLINICAL TRIAL: NCT00820625
Title: Ablation at St. Georg Hospital for Long-Standing Persistent Atrial Fibrillation - Pulmonary Vein Isolation With or Without Ablation of Complex Fragmented Atrial Potentials
Brief Title: Long-Standing Persistant Atrial Fibrillation-Pulmonary Vein Isolation With or Without Ablation
Acronym: Alster-Lost
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asklepios proresearch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1787; PV 2961 (Other: Ethical Board Hamburg)
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Atrial Fibrillation; Tachycardia
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ablation: pulmonary vein isolation
  Interventions: Procedure: pulmonary vein isolation
- 2 (Active Comparator): ablation: pulmonary vein isolation with additional ablation of fragmented potentials
  Interventions: Procedure: pulmonary vein isolation with additional ablation of fragmented potentials

INTERVENTIONS:
Procedure: pulmonary vein isolation — common pulmonary vein isolation procedure
  Arms: 1
Procedure: pulmonary vein isolation with additional ablation of fragmented potentials — common pulmonary vein isolation with additional but also common ablation of fragmented potentials
  Arms: 2

SUMMARY:
The chronic success rate, defined as freedom from any atrial tachyarrhythmias will increase from 35% to 60% by ablation of complex fragmented atrial electrograms potentials in addition to pulmonary vein isolation (PVI) as compared to PVI alone in patients with long-standing persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* long standing persistent atrial fibrillation > 6 months and < 5 years

Exclusion Criteria:

* renal failure
* left atrial size >55 mm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
data collection in view of acute and chronic success rate | 12 months

SECONDARY OUTCOMES:
data collection of complications in both groups and also procedure parameters | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, PhD, MD, Principal Investigator — Asklepios Klinik St. Georg, Department of Cardiology
Locations (1):
- Asklepios Klinik St. Georg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fink T, Schluter M, Heeger CH, Lemes C, Maurer T, Reissmann B, Riedl J, Rottner L, Santoro F, Schmidt B, Wohlmuth P, Mathew S, Sohns C, Ouyang F, Metzner A, Kuck KH. Stand-Alone Pulmonary Vein Isolation Versus Pulmonary Vein Isolation With Additional Substrate Modification as Index Ablation Procedures in Patients With Persistent and Long-Standing Persistent Atrial Fibrillation: The Randomized Alster-Lost-AF Trial (Ablation at St. Georg Hospital for Long-Standing Persistent Atrial Fibrillation). Circ Arrhythm Electrophysiol. 2017 Jul;10(7):e005114. doi: 10.1161/CIRCEP.117.005114. PMID 28687670